CLINICAL TRIAL: NCT00935181
Title: Respiratory Muscle Stretching in Patients With Chronic Obstructive Pulmonary Disease Submitted a Pulmonary Rehabilitation Program
Brief Title: Respiratory Muscle Stretching in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faculdade Evangelica do Parana (Other)
Responsible Party: Silvia Regina Valderramas, Faculdade Evangelica do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3145/06
Record Dates: First submitted 2009-06-29; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; diaphragm; muscle; stretching; exercises; dyspnea; respiratory muscle stretching; pulmonary rehabilitation; exercise training; improved exercise capacity, dyspnea, quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Dyspnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise training program (Experimental): The exercise training program consisted of three 90-minute sessions per week for eight weeks. Each session consisted of a stretching exercise, resistance that patients started at 70% of the initial one-repetition maximum (1RM: the maximum load which can be moved only once over the full range of motion without compensatory movements) in the first week (3x8 repetitions). Every week the load was increased by 5% of the 1RM, and endurance training (treadmill walking speed was set at 60% of the average speed obtained from the 6MWT (6MWTpeak) for 10 mins in the first week and was increased to 20 mins in week 8
  Interventions: Behavioral: respiratory muscle stretching

INTERVENTIONS:
Behavioral: respiratory muscle stretching — stretching exercises for respiratory muscles like diaphragm, pectoral, dorsalis etc
  Other Names: pulmonary rehabilitation

SUMMARY:
Objective: The investigators studied the effects of respiratory muscle stretching in an 8-week pulmonary rehabilitation program. Methods: This was a simple-blind parallel controlled trial, conducted an out-patient clinic. Twenty six patients with COPD (mean age 68 ± 6 y, percent of predicted FEV1 47 ± 16) were randomized to either respiratory muscle stretching group plus exercise training (RMS), and exercise training group (Sham), in an 8-week exercise program that had 3 sessions per week. The investigators measured inspiratory and expiratory muscle strength (by maximal inspiratory and expiratory pressure - PIM and PEM), exercise capacity (by 6-minute walk distance), dyspnea and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 40 and 75 years of age referred by a physician to the Pulmonary Rehabilitation Program
* With a clinical and spirometric diagnosis of moderate to severe COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD), in a stable condition (without exacerbations or infections for at least a month)
* Former smokers

Exclusion Criteria:

* Patients with a known history of asthma, or severe and/or unstable heart disease
* Any other pathological condition that could impair their physical activities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | 2 hours

SECONDARY OUTCOMES:
Exercise capacity | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R. Valderramas, Ph.D, Principal Investigator — Faculdade Evangelica do Paraná
Locations (1):
- Faculdade Evangelica do Paraná, Curitiba, Paraná, Brazil